CLINICAL TRIAL: NCT07349316
Title: The Effects of Weight Science and Nutrition Education on Weight Control Beliefs, Body Image, Self-Esteem and Eating Patterns in Undergraduate Dieters
Brief Title: The Effects of Weight and Nutrition Education on Weight Control Beliefs, Body Image, Self-Esteem and Eating Patterns in Undergraduate Dieters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Keisha Gobin, Co-Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19334
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Dietary Restraint
Keywords: Weight Control Beliefs; Dieters; Nutrition Counselling; Weight Science; Psychotherapeutic Interventions; Brief Intervention; Dietary Restraint
MeSH Terms: interventions — Nutrition Assessment; Diet, Healthy

STUDY DESIGN:
Intervention Model Description: This is an experimental study in which participants will be randomly assigned to one of three conditions: 1) weight science + control (sleep education); 2) control (sleep education) + healthy eating education; or 3) weight science + healthy eating education. The control component (sleep education) is the same in both Group 1 and Group 2 and is intended to serve as a pure placebo, not expected to influence the study's primary outcomes.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Weight Science Education and Sleep Education (Control) (Active Comparator): Participants in the Weight Science Education and Sleep Education (Control) arm will be receiving both those educational interventions after answering questionnaires. This arm assesses the hypothesis that weight science education alone will decrease belief in personal control over weight and will have little to no effect on belief in choosing a healthy lifestyle/weight acceptance.
  Interventions: Other: Weight Science Education; Other: Sleep Education
- Nutrition Education and Sleep Education (Control) (Active Comparator): Participants in the Nutrition Education and Sleep Education (Control) arm will be receiving both those educational interventions after answering questionnaires. This arm assesses the hypothesis that nutrition education alone will increase belief in choosing a healthy lifestyle or weight acceptance, but will have little to no effect on the belief in personal control over weight.
  Interventions: Other: Nutrition Education; Other: Sleep Education
- Weight Science Education and Nutrition Education (Experimental): Participants in the Weight Science Education and Healthy Eating Education arm will be receiving both those educational interventions after answering questionnaires. This arm assesses the main hypothesis that weight science and nutrition teaching combined will both decrease the belief of personal control over weight and an increase the belief in choosing a healthy lifestyle/weight acceptance.
  Interventions: Other: Weight Science Education; Other: Nutrition Education

INTERVENTIONS:
Other: Weight Science Education — The weight science educational video discusses the research on the genetic contribution to body weight; the role of genetics in how individuals' body weight responds to over-eating; the research comparing the efficacy of different dieting approaches; the research on the long-term efficacy of behavioural approaches to weight loss; weight loss in obesity; research on the weight-loss registry looking at successful weight losers; and research on weight control beliefs. The video is narrated by Dr. Michele Laliberte, a licensed clinical psychologist, and the information is consistent with current research and recommendations. There is no deception involved and it is made clear to participants that the information they are being provided is based on current research and the purpose is to understand the impact of this information on their attitudes and beliefs.
  Other Names: Weight Education; Weight Science
  Arms: Weight Science Education and Nutrition Education; Weight Science Education and Sleep Education (Control)
Other: Nutrition Education — The healthy nutrition educational video discusses the development of food guides around the world; a definition and description of benefits of the "basics" of healthy eating (e.g., regular eating, balanced eating and pleasurable eating); a review of the macronutrients and their importance to health; a review of the recommendations concerning the specific food groups in the Canada's food guide; and how to put this all together to create a healthy eating plan. The video is narrated by Dr. Michele Laliberte, a licensed clinical psychologist, and the information is consistent with current research and recommendations. There is no deception involved and it is made clear to participants that the information they are being provided is based on current research and the purpose is to understand the impact of this information on their attitudes and beliefs.
  Other Names: Healthy Eating Education; Healthy Eating; Healthy Nutrition Education
  Arms: Nutrition Education and Sleep Education (Control); Weight Science Education and Nutrition Education
Other: Sleep Education — The sleep hygiene educational video, which is an active control, reviews the cognitive, emotional, physical health and weight implications of good quality sleep; provides a review of good sleep hygiene; and provides an overview of how to manage insomnia. The video is narrated by Dr. Michele Laliberte, a licensed clinical psychologist, and the information is consistent with current research and recommendations. There is no deception involved and it is made clear to participants that the information they are being provided is based on current research and the purpose is to understand the impact of this information on their attitudes and beliefs.
  Other Names: Healthy Sleep; Healthy Sleep Education; Sleep Hygiene
  Arms: Nutrition Education and Sleep Education (Control); Weight Science Education and Sleep Education (Control)

SUMMARY:
People who diet typically believe they can control their weight. People who believe they should control their weight are more likely to have poor body image, low self-esteem and disordered eating. People who believe they should aim for a healthy lifestyle and accept their natural weight have better body image, better self-esteem and less disordered eating. This study will compare three types of education in undergraduate dieters. In the first, the investigators will teach how the body naturally controls weight. In the second, the investigators will teach about healthy eating. In the third, the investigators will teach about how the body naturally controls weight and healthy eating. The study is testing whether teaching about how the body naturally controls weight and healthy eating changes people's beliefs about weight. The study also tests whether changing people's beliefs about weight will change their body satisfaction, their feelings about themselves, and their intention to diet.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students at McMaster University
* Individuals who are restricting their eating to try and lose weight.
* Self-identified women
* Ages 18 or over
* Normal (or corrected to normal) hearing
* Normal (or corrected to normal) vision

Exclusion Criteria:

- Self-identified men

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in beliefs on the ability to control one's weight (weight control beliefs). | From baseline measure to the end of the intervention at approximately one hour.
  Decreased score on the Weight Control Beliefs questionnaire post-intervention compared to pre-intervention questionnaire score, where a total score of 17 is equivalent to beliefs that weight is not entirely under personal control and a total score of 68 indicates beliefs that weight is entirely under personal control.

SECONDARY OUTCOMES:
Change in restrained eating | From baseline measure to the end of the intervention at approximately one hour.
  Decreased score on the cognitive restraint subscale of the Three-Factor Eating Questionnaire Revised-18 (TFEQ-R18) post-intervention compared to pre-intervention questionnaire score. A cognitive restraint score of 24 is equivalent to high dietary restraint, and a cognitive restraint score of 6 indicates low dietary restraint.
Change in the intent to diet | From baseline measure to the end of the intervention at approximately one hour.
  Decreased mean score on the Dieting Intentions Scale (DIS) post-intervention compared to pre-intervention questionnaire score. A mean score of 7 is equivalent to a strong intent to diet, and a mean score of 1 indicates a low intent to diet.
Change in self-esteem | From baseline measure to the end of the intervention at approximately one hour.
  Increased score on the Rosenberg Self-Esteem scale (RSE) post-intervention compared to pre-intervention questionnaire score. A total score of 0 is equivalent to low self-esteem, and a total score of 30 indicates a high self-esteem.
Change in body appreciation | From baseline measure to the end of the intervention at approximately one hour.
  Increased score on the Body Appreciation Scale (BAS) post-intervention compared to pre-intervention questionnaire score. A score of 10 is equivalent to low body appreciation, and a score of 50 indicates high body appreciation.

OTHER OUTCOMES:
Change in disordered eating behaviours and attitudes | From baseline measure to the end of the intervention at approximately one hour.
  Decreased mean score on the Eating Disorders Examination Questionnaire 6.0 (EDE-Q6) post-intervention compared to pre-intervention questionnaire score. A mean score of 6 is equivalent to a high frequency and severity of behaviours associated with a diagnosis of an eating disorder, and a mean score of 0 indicates a low frequency and severity of behaviours associated with a diagnosis of an eating disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Participants are providing consent for inclusion in this singular study.

REFERENCES:
- [Background] Laliberte MM, Lucibello KM. Weight control beliefs in the treatment of binge-eating disorder: Why might they matter? Int J Eat Disord. 2022 Jun;55(6):820-825. doi: 10.1002/eat.23713. Epub 2022 Apr 7. PMID 35388511
- [Background] Laliberte, M. M., Balk, D., Tweed, S., Smith, J., & Ghai, A. (2014). The impact of education on weight control beliefs. Ethnicity and Inequalities in Health and Social Care, 7(2), 86-95. https://doi.org/10.1108/EIHSC-11-2013-0041
- [Background] Laliberte, M. M., Newton, M., McCabe, R., & Mills, J. S. (2007). Controlling Your Weight Versus Controlling Your Lifestyle: How Beliefs about Weight Control Affect Risk for Disordered Eating, 10534_2006_9060_Fig3_HTML.gif Dissatisfaction and Self-esteem. Cognitive Therapy and Research, 31(6), 853-869. https://doi.org/10.1007/s10608-006-9104-z

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT07349316/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT07349316/ICF_001.pdf